CLINICAL TRIAL: NCT01584973
Title: Changes in Inter-joint Coordination and Muscle Activation After Cruciate Ligament Injury of the Knee Joint
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201108032RC
Record Dates: First submitted 2012-04-24; First posted 2012-04-25 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-04

CONDITIONS: To Investigate the Change of Inter-joint Coordination and Muscle Activation in Patients With Cruciate Ligament Injury During Stair Negotiation.

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- cruciate ligament group
- control group

SUMMARY:
Stair negotiation is an important activity of daily living. Patients with cruciate ligament injury may have difficulty in stair negotiation because of the proprioception deficit and neuromuscular deficit caused by ligament injury. However, the influence of knee cruciate ligament injury on the control of movement is still unclear. Since inter-joint coordination can provide the information of relationship between angle position and angle velocity, it may be useful to analysis the change of movement pattern.This current study aimed to investigate the change of inter-joint coordination and muscle activation in patients with cruciate ligament injury during stair negotiation.

ELIGIBILITY:
Inclusion Criteria:

* unilateral cruciate ligament injury or unilateral cruciate ligament reconstructed after 3 month
* able to climb up and down with step-over-step pattern
* BMI within 18 to 30

Exclusion Criteria:

* complex ligament injury
* lower limb fracture in recent years
* meniscus injury
* systematic disorder which would affect the balance and ambulation

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: unilateral cruciate ligament injury or unilateral cruciate ligament reconstructed after 3 month
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2012-04

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Li Hsu, PhD, Principal Investigator — School of physical therapy, National Taiwan University
Locations (1):
- School & Graduate Institute of Physical Therapy, College of Medicine, National Taiwan University, Taipei, Taiwan